CLINICAL TRIAL: NCT01690585
Title: Efficacy of Parenteral Iron Supplementation After Gastrointestinal Bleeding in Subjects Over 65
Acronym: FerHem
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/123/HP
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Gastrointestinal Hemorrhage; Anemia
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferinject 1000 mg (Experimental): Intravenous Administration of 1000 mg of ferinject Volume of infusion : 250 mL
  Interventions: Drug: Ferinject 1000 mg
- Placebo (Placebo Comparator): Intravenous administration of 250 ml of sodium chlorure 0.9 %
  Interventions: Drug: Sodium chlorure 0,9 %

INTERVENTIONS:
Drug: Ferinject 1000 mg
  Arms: Ferinject 1000 mg
Drug: Sodium chlorure 0,9 %
  Arms: Placebo

SUMMARY:
The upper and lower gastrointestinal bleeding, not related to portal hypertension, is a common disorder in the elderly. Indeed, in 1996, in a French study, the median age of patients hospitalized for upper gastrointestinal bleeding was 68. During the same period in the studies reported in English the median age was 71. If epidemiological data concerning lower gastrointestinal bleeding are rare, the average age of hospitalized patients varies from 63 to 77 depending on the study. Due to improvement in endoscopic haemostatic procedures and current resuscitation methods, gastrointestinal bleeding prognosis has greatly improved, whereas anaemia related to a bleeding episode remains a frequent complication of gastrointestinal bleeding in elderly patients.

Among elderly patients over 65, the prevalence of anaemia varies from 8 to 44% depending on the criteria used and populations studied. The occurrence of a bleeding episode can either induce anaemia or exacerbate pre-existing anaemia. Physicians in charge of gastrointestinal bleeding are often unaware of anaemic consequences in the elderly patients which can often be serious. Various studies have shown that anaemia increases morbidity and mortality rates in the elderly. Life expectancy is independently significantly lower for anaemic patients over 65, than for non-anaemic subjects. Anaemia is also a risk factor for the occurrence of cardiovascular and neurological complications, impairment in cognitive function and increased risk of falling.

Iron deficiency and anaemia induced by bleeding episodes in patients over 65 hospitalized for upper or lower gastrointestinal bleeding should be corrected rapidly and effectively. Currently, the cost and risks of infection or cardiovascular-related complications of transfusions lead to limiting red blood cell transfusion with a goal average of 9 g/dL haemoglobin. It is also necessary to develop alternatives to massive transfusions. The correction of iron deficiency promotes erythropoiesis and can quickly correct anaemia.

In clinical practice, the effectiveness of iron intake by the oral route is limited by the frequent occurrence of significant gastrointestinal side effects that limit patient compliance and limited absorption necessitating prolonged treatment to correct iron deficiency.

The black colour of stools caused by taking oral iron supplements also makes it difficult to detect a possible recurrence of bleeding after hospitalization.

The prescription of intravenous iron seems more suitable for a rapid and complete correction of iron deficiency after gastrointestinal bleeding. The main objective of our study is to evaluate efficacy of intravenous iron for the correction of anaemia, measured by haemoglobin at week 6 (W6) in patients aged over 65, after gastrointestinal bleeding. Secondary objectives were to assess the speed of anaemia correction, the tolerance of intravenous iron supplementation, the rate of re-hospitalization within 6 months after discharge and patients quality of life. This is a prospective multicenter randomized study versus placebo. After obtaining informed consent, all patients aged over 65 admitted with upper or lower gastrointestinal bleeding, with successful outcome, not related to portal hypertension, responsible for persistent anaemia (definition: Hb < 11 g / dL) after hospitalization will be included in the study. Patients will be treated for their bleeding event in the usual manner of each centre with target for transfusion of 9 g / dL haemoglobin. The absence of external bleeding and haematocrit and/or constant haemoglobin levels will be considered as the end of bleeding.

Day 1 was arbitrarily defined as the day the patient left hospital. The protocol at Day - 1 included: obtaining informed consent of the patient, determination of iron and ferritin blood levels and complete blood count. and randomization intravenous iron injection , (Ferinject) versus Placebo. Intravenous iron injection will be performed at Day 0. A complete blood count will be performed at week 6 and month 6. Patients will be reviewed in consultation at week 6 and at month 6 to obtain related intercurrent events and assess their quality of life.

The results of this study could lead to changes in the care of older patients hospitalized for gastrointestinal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 65 hospitalized for upper or lower GI bleeding with positve outcome during hospitalization without surgery, and with persistent anaemia (Hb <11g/dL),
2. Signed informed consent,
3. Patients with National Health Insurance,

Exclusion Criteria:

1. Uncontrolled haemorrhage defined by any new externalizing and / or a decrease of haemoglobin and haematocrit levels,
2. GI bleeding related to portal hypertension or malignancy,
3. The absence of anaemia,
4. Cancer evolution,
5. Patient under guardianship, curatorship or unable to supply consent,
6. Iron overload,
7. History of asthma
8. History of eczema
9. Hypersensitivity to any component
10. Decompensated liver cirrhosis
11. Infection during treatment or uncontrolled infection 12 Rheumatoid arthritis

13. Acute renal failure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Haemoglobin level | Week 6

SECONDARY OUTCOMES:
Assessment of the tolerance of intravenous iron supplementation | Day 0
  Number of Adverse Event (AE) and Serious Adverse Event(SAE) occurence.
Assessment of the tolerance of intravenous iron supplementation | Week 6
  Number of Adverse Event (AE) and Serious Adverse Event(SAE) occurence.
re-hospitalization rate | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SAVOYE, Pr, Principal Investigator — UH Rouen
Locations (13):
- France (13):
  - CHU d'Amiens, Amiens
  - CHU de Caen, Caen
  - CH de Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CHI le Raincy Montfermeil, Le Raincy
  - CH de Montélimar, Montélimar
  - GH du havre, Montivilliers
  - CHU de Nice, Nice
  - CH d'Orléans, Orléans
  - CHU de Pau, Pau
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CH de Valenciennes, Valenciennes

REFERENCES:
- [Derived] Richard N, Arab-Hocine N, Vannier M, Leblanc-Boubchir R, Pelaquier A, Boruchowicz A, Musikas M, Amil M, Fumery M, Nahon S, Arotcarena R, Gelsi E, Maurin A, Hebuterne X, Savoye G. Efficacy of ferric carboxymaltose on haemoglobin response among older patients with gastrointestinal bleeding: a randomised clinical trial. Age Ageing. 2024 May 1;53(5):afae085. doi: 10.1093/ageing/afae085. PMID 38706390